CLINICAL TRIAL: NCT06592144
Title: TESTO-TRIAL: Randomized Clinical Trial on the Use of Testosterone in Critically Ill Patients
Brief Title: TESTO-TRIAL: Use of Testosterone in Critically Ill Patients
Acronym: TT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leticia Maria Defendi Barboza Marson (Other)
Responsible Party: Sponsor-Investigator, Leticia Maria Defendi Barboza Marson, PhD student, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CAAE76790723.5.0000.5440072024
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Weaning Failure; Muscle Weakness; Mechanical Ventilation Complication; ICU Acquired Weakness; Mobility Limitation
Keywords: Testosterone; Mechanical ventilation; Weaning; Critical Illness
MeSH Terms: conditions — Muscle Weakness; Mobility Limitation; Critical Illness | interventions — testosterone 17 beta-cypionate; Sesame Oil

STUDY DESIGN:
Intervention Model Description: Intervention Group: Participants will receive 200 mg of testosterone cypionate intramuscularly every 5 days, up to a maximum of 3 doses.
  Control Group: Participants will receive sesame oil (placebo) intramuscularly every 5 days, up to a maximum of 3 doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All assistant team members (physicians, pharmacists, nurses, etc.) and statisticians responsible for the analyses will remain blind to the identity of the treatments throughout the study.
  The placebo (sesame oil) will be prepared in a similar packaging and with a volume identical to that of testosterone cypionate.
  If a patient experiences an adverse effect potentially related to the medication, the attending physician may request to break the study blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Experimental): Participants will receive 200 mg of testosterone cypionate intramuscularly every 5 days, up to a maximum of 3 doses.
  Interventions: Drug: Testosterone cypionate (200mg/3ml)
- Sesame oil (Placebo Comparator): Participants will receive sesame oil (placebo) intramuscularly every 5 days, up to a maximum of 3 doses.
  Interventions: Other: Sesame oil (3ml)

INTERVENTIONS:
Drug: Testosterone cypionate (200mg/3ml) — It will be administered intramuscularly every 5 days, totaling 3 doses.
  Arms: Testosterone
Other: Sesame oil (3ml) — It will be administered intramuscularly every 5 days, totaling 3 doses.
  Arms: Sesame oil

SUMMARY:
The objective of this study is to evaluate whether the use of the anabolic agent testosterone cypionate in critically ill patients, compared to placebo, increases the number of ventilator-free days

DETAILED DESCRIPTION:
It will be a randomized, controlled, double-blind, single-center clinical trial conducted in the Intensive Care Unit (ICU) of the State Hospital of Serrana (HE Serrana). Patients admitted to the ICU who meet the eligibility criteria and have given written informed consent will be randomized into control and intervention groups. Forty-seven patients will be included in each group, totaling 94 patients. The intervention group will receive 200 mg of testosterone cypionate intramuscularly every 5 days for a total of 3 doses. The control group will receive a placebo on the same schedule. After inclusion in the study, demographic and clinical data, laboratory results, ultrasonographic measurements, and functionality and muscle strength scores will be assessed on days 1, 5, 10, and 15 in the ICU and until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation (MV) for seven days or more, or patients on MV with an unsuccessful weaning attempt for at least three days. An unsuccessful weaning attempt is defined as the patient undergoing a Spontaneous Breathing Trial (SBT) on three different days without success, according to the ICU protocol;
* Over 18 years old;
* Patients with optimized nutritional therapy, defined by caloric and protein goals met for at least three days;
* Signing the informed consent form (ICF).

Exclusion Criteria:

* Hypersensitivity to the medication, the vehicle of the medication, or the placebo (sesame oil);
* Venous or arterial thrombosis in the past six months, including acute myocardial infarction, ischemic stroke, acute arterial occlusion, mesenteric ischemia, venous thromboembolism, or pulmonary embolism;
* Left Ventricular Ejection Fraction (LVEF) below 35%;
* Glutamic-pyruvic transaminase/Alanine Aminotransferase (GPT/ALT) greater than five times the normal level and impaired bilirubin excretion;
* Patients with liver cirrhosis (CHILD > B);
* Pregnant or lactating women;
* Women of childbearing age;
* Hematocrit >52%;
* Refractory shock, defined as requiring a norepinephrine dose > 0.5 mcg/kg/min or a vasopressin dose > 0.04 IU/min;
* Thrombocytopenia < 20,000/mm³ without a transfusion plan;
* Personal history of prostate or breast cancer;
* Active neoplasm of any site;
* Primary neuromuscular disease, including Amyotrophic Lateral Sclerosis (ALS), Duchenne muscular dystrophy, myasthenia gravis, or Guillain-Barré syndrome;
* Current or previous spinal cord injury above C4 (tetraplegia);
* Patients with total limitation of therapeutic measures;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days at 28 days, starting from the date of randomization. | 28 days
  Evaluate whether the use of the anabolic steroid testosterone cypionate, compared to a placebo, increases the number of ventilator-free days in critically ill patients.

SECONDARY OUTCOMES:
Length of stay in the hospital, measured in days. | ICU and hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on the length of hospital stays.
Length of stay in the ICU, measured in days. | ICU and hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on the length of ICU (Intensive Care Unit) stays.
Ventilator weaning time in days, starting from the date of randomization. | ICU stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on the duration of mechanical ventilation.
In-hospital mortality from any cause. | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on in-hospital mortality.
Sequential Organ Failure Assessment (SOFA) score during the ICU stay, starting from the date of randomization. | ICU stay, assessed up to 8 weeks.
  Evaluate the effects of using testosterone cypionate on the SOFA score during ICU hospitalization. This score is used to assess the degree of organ dysfunction in the patient, with scores ranging from 0 to 24 points; the higher the score, the greater the severity and risk of mortality in critically ill patients.
Diaphragmatic muscle thickness. | Hospital stay, assessed up to 8 weeks
  Evaluate the effects of using testosterone cypionate on the diaphragmatic muscle during hospitalization by measuring diaphragm thickness (in millimeters) through ultrasonography.
Diaphragmatic thickening fraction. | Hospital stay, assessed up to 8 weeks
  Evaluate the effects of using testosterone cypionate on the diaphragmatic muscle during hospitalization through ultrasonography. The thickening fraction is calculated using the following equation: (Final inspiratory diaphragm thickness - Final expiratory diaphragm thickness)/Final expiratory diaphragm thickness × 100. If the result is greater than 36%, it predicts successful weaning from mechanical ventilation.
Skeletal muscle assessment: quadriceps thickness. | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of using testosterone cypionate on the thickness of the rectus femoris muscle by measuring its thickness at maximum and minimum compression through ultrasonographic analysis.
Skeletal muscle assessment: Medical Research Council Sum-Score (MRC-SS). | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate on muscle strength gain using the MRC, which scores muscle strength from 0 (no contraction) to 5 (normal muscle contraction) for shoulder flexors, elbow flexors, wrist extensors, hip flexors, knee extensors, and ankle dorsiflexors, totaling 60 points.
Skeletal muscle assessment: dynamometry. | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone on muscle strength gain by measuring handgrip strength using dynamometry with the JAMAR dynamometer.
Skeletal muscle assessment: calf circumference. | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone on muscle mass gain indirectly by measuring calf circumference (in centimeters).
Functionality and quality of life of critically ill patients during hospital stay: ICU Mobility Scale. | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on functionality scores, including the ICU Mobility Scale (IMS) to objectively measure the mobility of patients in the ICU. This scale has a score ranging from 0 to 10, where a score of zero indicates low mobility (interpreted as a patient who only performs passive bed exercises) and a score of 10 indicates high mobility (interpreted as a patient who is independently ambulatory, without assistance).
Functionality and quality of life of critically ill patients during hospital stay: Perme Intensive Care Unit Mobility Score. | Hospital stay, assessed up to 8 weeks.
  Perme Intensive Care Unit Mobility Score objectively measures the mobility condition of a patient in the ICU. This mobility scale has a score ranging from 0 to 32 points, divided into 15 items grouped into 7 categories: mental state, potential barriers to mobility, functional strength, bed mobility, transfers, assistive devices for ambulation, and endurance measures. In this scale, a higher score indicates greater mobility and less need for assistance. Conversely, a lower score indicates reduced mobility and a greater need for assistance.
Functionality and quality of life of critically ill patients during hospital stay: FSS-ICU (Functional Status Score for the Intensive Care Unit). | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone on the functionality of critically ill patients using the FSS-ICU, a tool that involves five functional tasks (rolling, transferring from supine to sitting, transferring from sitting to standing, sitting on the edge of the bed, and walking). Each task is assessed using an 8-point ordinal scale, ranging from 0 (completely unable to perform) to 7 (complete independence).
Functionality and quality of life of critically ill patients during hospital stay: TUG (Timed Up and Go). | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on functionality scores, including the TUG (Timed Up and Go). The parameter evaluated is the time spent (in seconds) to rise from a chair, walk a distance of 3 meters, and return to sit down. The test is considered normal when the time taken is less than 10 seconds. If the time is between 10 and 19 seconds, the elderly person is considered to have a moderate risk of falling, and this risk increases when the time is 20 seconds or more.
Correlation of serum testosterone levels, clinical characteristics, and demographics of patients. | Hospital stay, assessed up to 8 weeks.
  Evaluate the correlation between patients clinical and demographic characteristics, as well as free testosterone serum levels in the placebo and intervention groups.
Correlation with serum levels of hemoglobin and hematocrit, in addition to patients clinical characteristics. | Hospital stay, assessed up to 8 weeks.
  Evaluate the correlation between patients clinical and demographic characteristics and laboratory test levels, about the use of testosterone and the stimulation of erythropoietin production, leading to an increase in red blood cell production and, consequently, an increase in hemoglobin (normal value: 12.5 to 17.2 g/dL) and hematocrit (37-49%).
Correlation with serum albumin levels and patients clinical characteristics. | Hospital stay, assessed up to 8 weeks.
  Evaluate the correlation between patients clinical and demographic characteristics and laboratory test levels, considering the affinity of total testosterone to albumin (normal value: 3.2 to 4.8 g/dL).
Functionality and quality of life of critically ill patients during hospital stay: the Barthel Index. | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of using testosterone cypionate on functionality scores, including the Barthel Index at hospital discharge. The Barthel Index consists of ten items, such as feeding, transferring from bed to chair and back, personal hygiene, using the toilet, bathing, walking on a flat surface, stairs, dressing, fecal continence, and bladder continence. Each item has variable scores ranging from zero to fifteen points, depending on the individuals level of functional dependence. The maximum score is 100, which is assigned only if the patient does not require any assistance.
Quality of life of critically ill patients during hospital stay: EQ-5D (EuroQol 5-Dimension). | Hospital stay, assessed up to 8 weeks.
  Evaluate the effects of testosterone cypionate use on quality of life, including the EQ-5D (EuroQol 5-Dimension) at hospital discharge.
  The EQ-5D includes five levels of response for each of the five variables assessed: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each variable is scored from 1 to 5, where 1 indicates no problems and 5 indicates extreme problems. The final score is a combination of the numbers assigned to each variable, resulting in a five-digit code that represents the patients health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Estadual Serrana, Serrana, SP/Brazil, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participant data will be available upon completion of clinical trials and publication of the results of the completed study upon request to the corresponding author. Proposals will be reviewed and approved by the sponsor, researcher, and staff on the basis of scientific merit and absence of competing interests. After the proposal has been approved, data can only be shared through a secure online platform after data access code exchange and a confidentiality agreement are signed.

REFERENCES:
- [Background] Wischmeyer PE, Suman OE, Kozar R, Wolf SE, Molinger J, Pastva AM. Role of anabolic testosterone agents and structured exercise to promote recovery in ICU survivors. Curr Opin Crit Care. 2020 Oct;26(5):508-515. doi: 10.1097/MCC.0000000000000757. PMID 32773614
- [Background] Stanojcic M, Finnerty CC, Jeschke MG. Anabolic and anticatabolic agents in critical care. Curr Opin Crit Care. 2016 Aug;22(4):325-31. doi: 10.1097/MCC.0000000000000330. PMID 27272101
- [Background] Anstey MH, Rauniyar R, Fitzclarence E, Tran N, Osnain E, Mammana B, Jacques A, Palmer RN, Chapman A, Wibrow B. Muscle Growth and Anabolism in Intensive Care Survivors (GAINS) trial: a pilot randomised controlled trial. Acute Crit Care. 2022 Aug;37(3):295-302. doi: 10.4266/acc.2021.01767. Epub 2022 Jun 27. PMID 35791659
- [Background] Basaria S, Coviello AD, Travison TG, Storer TW, Farwell WR, Jette AM, Eder R, Tennstedt S, Ulloor J, Zhang A, Choong K, Lakshman KM, Mazer NA, Miciek R, Krasnoff J, Elmi A, Knapp PE, Brooks B, Appleman E, Aggarwal S, Bhasin G, Hede-Brierley L, Bhatia A, Collins L, LeBrasseur N, Fiore LD, Bhasin S. Adverse events associated with testosterone administration. N Engl J Med. 2010 Jul 8;363(2):109-22. doi: 10.1056/NEJMoa1000485. Epub 2010 Jun 30. PMID 20592293
- [Background] Anstey M, Desai S, Torre L, Wibrow B, Seet J, Osnain E. Anabolic Steroid Use for Weight and Strength Gain in Critically Ill Patients: A Case Series and Review of the Literature. Case Rep Crit Care. 2018 May 7;2018:4545623. doi: 10.1155/2018/4545623. eCollection 2018. PMID 29854477
- [Background] Li H, Guo Y, Yang Z, Roy M, Guo Q. The efficacy and safety of oxandrolone treatment for patients with severe burns: A systematic review and meta-analysis. Burns. 2016 Jun;42(4):717-27. doi: 10.1016/j.burns.2015.08.023. Epub 2015 Oct 9. PMID 26454425
- [Background] Dres M, Demoule A. Diaphragm dysfunction during weaning from mechanical ventilation: an underestimated phenomenon with clinical implications. Crit Care. 2018 Mar 20;22(1):73. doi: 10.1186/s13054-018-1992-2. PMID 29558983
- [Background] Zambon M, Greco M, Bocchino S, Cabrini L, Beccaria PF, Zangrillo A. Assessment of diaphragmatic dysfunction in the critically ill patient with ultrasound: a systematic review. Intensive Care Med. 2017 Jan;43(1):29-38. doi: 10.1007/s00134-016-4524-z. Epub 2016 Sep 12. PMID 27620292
- [Background] Haaksma ME, Smit JM, Boussuges A, Demoule A, Dres M, Ferrari G, Formenti P, Goligher EC, Heunks L, Lim EHT, Mokkink LB, Soilemezi E, Shi Z, Umbrello M, Vetrugno L, Vivier E, Xu L, Zambon M, Tuinman PR. EXpert consensus On Diaphragm UltraSonography in the critically ill (EXODUS): a Delphi consensus statement on the measurement of diaphragm ultrasound-derived parameters in a critical care setting. Crit Care. 2022 Apr 8;26(1):99. doi: 10.1186/s13054-022-03975-5. PMID 35395861
- [Background] Santana PV, Cardenas LZ, Albuquerque ALP, Carvalho CRR, Caruso P. Diaphragmatic ultrasound: a review of its methodological aspects and clinical uses. J Bras Pneumol. 2020 Nov 20;46(6):e20200064. doi: 10.36416/1806-3756/e20200064. eCollection 2020. PMID 33237154
- [Background] Santangelo E, Mongodi S, Bouhemad B, Mojoli F. The weaning from mechanical ventilation: a comprehensive ultrasound approach. Curr Opin Crit Care. 2022 Jun 1;28(3):322-330. doi: 10.1097/MCC.0000000000000941. PMID 35653254
- [Background] Galindo Martin CA, Monares Zepeda E, Lescas Mendez OA. Bedside Ultrasound Measurement of Rectus Femoris: A Tutorial for the Nutrition Support Clinician. J Nutr Metab. 2017;2017:2767232. doi: 10.1155/2017/2767232. Epub 2017 Mar 13. PMID 28386479
- [Background] Paris MT, Mourtzakis M, Day A, Leung R, Watharkar S, Kozar R, Earthman C, Kuchnia A, Dhaliwal R, Moisey L, Compher C, Martin N, Nicolo M, White T, Roosevelt H, Peterson S, Heyland DK. Validation of Bedside Ultrasound of Muscle Layer Thickness of the Quadriceps in the Critically Ill Patient (VALIDUM Study). JPEN J Parenter Enteral Nutr. 2017 Feb;41(2):171-180. doi: 10.1177/0148607116637852. Epub 2016 Jul 11. PMID 26962061
- [Background] Pardo E, El Behi H, Boizeau P, Verdonk F, Alberti C, Lescot T. Reliability of ultrasound measurements of quadriceps muscle thickness in critically ill patients. BMC Anesthesiol. 2018 Dec 27;18(1):205. doi: 10.1186/s12871-018-0647-9. PMID 30591032